CLINICAL TRIAL: NCT05635292
Title: Addressing Disability Effectively With Psychosocial Telemedicine (ADEPT Study): An Open-label, Multicenter Pragmatic Randomized Control Trial
Brief Title: Addressing Disability Effectively With Psychosocial Telemedicine
Acronym: ADEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 851901
Record Dates: First submitted 2022-11-10; First posted 2022-12-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-CBT (Experimental)
  Interventions: Behavioral: Tele-CBT
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Tele-CBT — 8 weekly 1-hr telemedicine visits with a licensed Ph.D. psychologist from the University of Pennsylvania (permissible to practice across state lines under PSYPACT), plus usual care and referral to an IBD Help Center (email, phone, online chat with IBD information specialist)
  Arms: Tele-CBT

SUMMARY:
This multi-site study will be implemented at 5 gastroenterology practices to recruit 420 adults with IBD to complete a baseline survey and enroll those with higher scores on a validated IBD-disability scale into a randomized controlled trial of telehealth-delivered cognitive behavioral therapy with a licensed psychologist versus usual care. The investigators aim to lay the foundations that will shift the paradigm of IBD clinical practice towards a new horizon of holistic and equitable high-value care.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old with a diagnosis of Crohn's disease (CD) or ulcerative colitis (UC)
2. Willingness to complete the baseline survey online. Participants in Aim 1 with moderate-to-severe disability based on the IBD Disability Index (IBD-DI) will be invited to the Aim 2 clinical trial
3. Able to consent and complete surveys in English.

Exclusion Criteria:

1. no/low disability (IBD-DI <35) on the baseline survey
2. inability or unwillingness to participate in telemedicine with a therapist
3. Have an existing relationship with a mental health specialist within the past 3 months
4. Lack of access to a computer, working internet connection, and a private environment to complete teletherapy sessions if they are randomized to this intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in the IBD Disability Index | 8 weeks
  Change in the IBD Disability is estimated by the 14-item validated IBD Disability Index (IBD-DI) in the intervention group (telemedicine-delivered psychosocial care) vs control group (usual care) in patients with moderate-to-severe baseline IBD-related disability pre and post intervention (week 0 and week 8). Total score ranges from 0-100, interpreted as 0-20 (no disability), 20-35 (mild disability), 35-50 (moderate disability), and 50-100 (severe disability).

SECONDARY OUTCOMES:
Cost-benefits of telemedicine-delivered psychosocial care | 8 weeks
  The cost-benefits of tele-CBT are estimated by 5-item validated Centers for Medicare & Medicaid Services (CMS)-certified FAIR Health database questionnaire titled the Treatment Inventory of Costs in Patients (TIC-P). The minimum value is $0, with no maximum value. Higher costs indicate worse outcome. In order to calculate the costs of productivity losses, the healthcare utilization encounter are multiplied by the cost price per unit. The cost of unpaid productivity loss is calculated by multiplying the productivity losses by a standard hourly rate for household care.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Sang Tse, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Tse CS, Hunt MG, Brown LA, Lewis JD. Inflammatory Bowel Diseases-related Disability: Risk Factors, Outcomes, and Interventions. Inflamm Bowel Dis. 2024 Mar 1;30(3):501-507. doi: 10.1093/ibd/izad182. PMID 37603844
- [Derived] Tse CS, Lewis JD, Horst SN, Saha S, Taleban S, Shah SA, Lutz M, Fiske HW, Brown LA, Kuehnel R, Bonhomme B, Weng CH, Weaver SA, Cross RK, Hunt MG; Crohn's and Colitis Foundation's Clinical Research Alliance. Inflammatory Bowel Diseases-Specific Cognitive Behavioral Therapy Delivered Through Telehealth Reduces Disability: Addressing Disability Effectively With Psychosocial Telemedicine Pragmatic Randomized Controlled Trial. Am J Gastroenterol. 2025 Jul 30. doi: 10.14309/ajg.0000000000003681. Online ahead of print. PMID 40736700
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Hunt M, Tse CS, Suh L, Yang E, Bui C, Davis A, Siddiqi R, Tian V. Psychotherapy process variables in implementation of CBT for inflammatory bowel disease:Therapist competence, fidelity, and patient themes. Behav Res Ther. 2025 Mar;186:104702. doi: 10.1016/j.brat.2025.104702. Epub 2025 Jan 31. PMID 39919362